CLINICAL TRIAL: NCT00517647
Title: Atomoxetine Pilot Study in Preschool Children With ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC04-22
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; atomoxetine; preschool children; efficacy; safety
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ATMX — Medication phase: After screening assessments are completed, the child will enter the medication phase of the study. The child will be started on atomoxetine at 0.5 mg/kg/day, with the dosage increased to a maximum dose of 1.8 mg/kg/day. The dose will be determined by how well the child responds to and tolerates the drug. The dose will be given twice a day to minimize side effects. After the optimum dose is determined, the child will be kept at this stable dose for 4 weeks.

SUMMARY:
The purpose of this study is to determine if atomoxetine (a common brand name is Strattera), a medicine that is used for treating older children with Attention Deficit and Hyperactivity Disorder (ADHD), is also safe and helpful for ADHD problems in young children. While atomoxetine is not approved by the FDA for use in children younger than 6 years, the FDA has given permission to study this drug in this age group.

DETAILED DESCRIPTION:
Prevalence of Attention Deficit Hyperactivity Disorder ADHD in school age children is estimated to be 2% to 11%. Many preschool age children have problems with hyperactivity, short attention span, impulsivity and other behavior dyscontrol and are quite likely to continue to have difficulties in elementary school years. Many of these children are referred for diagnosis and management of their difficult behavior and are diagnosed with ADHD. Children with ADHD often display disruptive behaviors that interfere with their functioning at school, home and in the community due to symptoms of hyperactivity, impulsiveness and inattention.

Symptoms of ADHD may be underdiagnosed and undertreated in preschool children. Preschool children with ADHD often require vigilant monitoring and supervision to ensure their safety. Symptoms of impulsivity, hyperactivity and distractibility often limit the effectiveness of educational and behavioral interventions. Hence, it is important to treat the symptoms of ADHD in children at an early age. Early intervention in children with ADHD may have an impact in the course of illness by abating longer-term disability in vulnerable children.

Pharmacological agents are considered a standard treatment recommendation in children with ADHD. Recently, a non-stimulant pharmacological agent, atomoxetine (ATMX), has been reported to be effective and safe in school-age children with ADHD. Data are not available for the usefulness of ATMX in children younger than 6 years. However, parents of younger children with ADHD are frequently asking practicing physicians to prescribe ATMX for their child since they do not want their child taking stimulants.

There is a need to carry out treatment trials with ATMX in preschool children with ADHD in order to collect data on how effective the drug is, its safety, and the best doses to administer to children with ADHD. Therefore, this study will be a pilot project to obtain preliminary data that will then be used to help set up a larger study that will examine preschool children with ADHD.

All subjects will be screened for eligibility inclusion and exclusion criteria. Since other therapies including behavior therapy are routinely indicated, for ethical reasons subjects will continue to receive all concurrent therapies throughout the study period. All concurrent therapies will be stabilized for a minimum period of 2 weeks prior to the child's entry into the drug phase of the study. At each medication follow-up visit, a detailed history will be obtained and recorded for all concurrent treatments.

If a child enrolls in this study, his/her participation will last approximately 7 to 13 weeks with a minimum of 7 outpatient daytime visits. The visits will be weekly in the beginning and then every other week once the child is taking an optimum dose of atomoxetine. Visits will take 1-5 hours each and will take place at the Department of Psychiatry in the Arizona Health Sciences Center (Tucson). The study consists of 2 periods.

Screening assessment: The screening visit(s) is/are used to determine if a child is eligible for participation. The child's teacher/daycare provider (with the parent's permission) and the parent(s) will need to complete some forms describing the child's problems with overactivity, impulsivity and inattention. The screening assessments may be completed over 1-2 visits. Each visit will take about 3-5 hours to complete. The research staff will evaluate each child to see if s/he has ADHD. Parents will be interviewed about their child's behavior. The child's teacher will be given several rating forms to complete. Parents will be asked to complete some questions about their child's development. Both parents (if available) and will be interviewed about their family histories.

After it is determined that a child is eligible to participate, there will be a baseline visit. The child's previous ineffective medication will be discontinued. The ratings done at the first visit will be repeated, including both the teacher and parent rating scales. The child will have vital signs taken including height, weight, blood pressure and pulse rate, an electrocardiogram (EKG) (a test of heart rhythm recorded by putting sticky pads on the chest), a urine test and a blood test (about 10cc or 1 tablespoon). The doctor will ask the parents about the child's medical history. Parents will be told about any abnormal laboratory values or physical findings that may be discovered during this study. This information will also be available to the child's pediatrician if the parents request this be done.

Medication phase: After screening assessments are completed, the child will enter the medication phase of the study. The child will be started on atomoxetine at 0.5 mg/kg/day, with the dosage increased to a maximum dose of 1.8 mg/kg/day. The dose will be determined by how well the child responds to and tolerates the drug. The dose will be given twice a day to minimize side effects. After the optimum dose is determined, the child will be kept at this stable dose for 4 weeks.

At each visit, vital signs will be taken including height, weight, blood pressure, and pulse rate. Interviews, play assessments, checklist, and questionnaires will be completed at each visit in order to assess how well the child is doing, and whether there are symptoms or side effects. Teachers will also continue to be asked to fill out assessments.

If the child's behavior gets worse or s/he experiences any side effects, parents should call the study doctor immediately and it will be determined if any changes in the child's treatment will need to be made. Participants will be given a card with telephone numbers and important information needed to get in touch with the doctor at any time, day or night.

Some of the screening assessments will be videotaped/audiotaped. These tapes will be used for later coding, supervision of the child's doctor/therapist, review by offsite consultants/mentors, training of other doctors/therapists, and/or for presentations at conferences. The tapes can be erased at any time during or after the session at the parent's request.

ELIGIBILITY:
Inclusion Criteria:

* Child must be 36-69 months old at the time of screening to insure that the child can complete the short-term safety and efficacy trial before the age of 6 years.
* Child must have categorical and dimensional evidence of clinically significant ADHD symptoms in multiple settings that have been present for at least six months.
* ADHD symptoms must cause significant functional impairment in the child. Child must meet impairment scale threshold based on Children's Global Assessment Scale (C-GAS, Shaffer, Gould, Brasic et al., 1983) score < 60.
* Child must have resided with primary caretaker for at least 6 months prior to the screening.
* Child's heart rate must be within the 98th percentile and blood pressure within the 95th percentile by age and gender and oral temperature values within the normal range.

Exclusion Criteria:

* Child with prior failed treatment with an adequate trial of ATMX (defined by a minimum of 1.8 mg/kg/day for 4 weeks) or known hypersensitivity to ATMX. Prior failure on stimulants or other psychotropics will not be the sole reason for exclusion.
* Child is taking MAOI or there have been less than 2 weeks since it was discontinued.
* Concurrent treatment with other medications that have CNS effects or that affect performance (e.g., antidepressants, antipsychotics, alpha-agonists, adrenergic blockers, lithium carbonate, sedating antihistamines, decongestant or sympathomimetics). Child should be off of previous psychotropic medications for a minimum duration of one week for stimulants, clonidine or guanfacine; two weeks for bupropion, tricyclic antidepressants, venlafaxine, SSRIs (except fluoxetine and citalopram), valproate; and three weeks for fluoxetine, citalopram, and neuroleptics.
* Child has narrow angle glaucoma.
* Child who has a major medical condition that would interfere with involvement in the study or would be affected negatively by ATMX (i.e., heart disease, high blood pressure, glaucoma, untreated or unstable hyperthyroidism, uncontrolled seizure disorder, or illnesses that would require hospitalization).
* Child with co-morbid psychiatric diagnoses of Major Depression, Bipolar Disorder, a psychotic disorder, or other psychiatric disorders in addition to ADHD that requires concurrent treatment with additional/alternative medication.
* Current history of physical, sexual, or emotional abuse.
* The patient has taken an investigational drug within the last 30 days.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2004-04; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
A reduction of 30% in the Hyperactive-Impulsive (HI) subscale scores of the Conners Rating Scale-Revised, which indicates an improvement in both efficacy and a significant clinical improvement in the child. | 7 to 13 weeks

SECONDARY OUTCOMES:
Decrease in ADHD specific symptom severity and impairment | 7 to 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jaswinder K Ghuman, M.D., Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Department of Psychiatry, Tucson, Arizona, United States